CLINICAL TRIAL: NCT05877703
Title: Effects of Open Versus Close Kinetic Chain Exercise Training Program With Lifestyle Modification and Patient's Education in Grade 3 Knee Osteoarthritis
Brief Title: Open Versus Close Chain Exercise Effects With Lifestyle Modification and Education in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0103
Record Dates: First submitted 2023-05-18; First posted 2023-05-26 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: close kinetic chain exercises (Experimental): Group A will be treated with close kinetic chain exercises including static cycling with lifestyle modification and patient's education including quadriceps drill with lifestyle modification and patient's education about 30 minutes per session including 10 min of walking as a warm up for total duration of 12 weeks with 3 sessions per week. Assessment will be done by therapist at 0 week, 4 weeks, 8 weeks and 12 weeks
  Interventions: Other: close kinetic chain exercises
- Group B: open kinetic chain exercises (Active Comparator): Group B will be treated with open kinetic chain exercises including quadriceps drill with lifestyle modification and patient's education about 30 minutes per session including 10 min of walking as a warm up for total duration of 12 weeks with 3 sessions per week. Group B performed scar mobilization exercises only for 3 weeks. Assessment will be done by therapist at 0 week, 4 weeks, 8 weeks and 12 weeks
  Interventions: Other: open kinetic chain exercises

INTERVENTIONS:
Other: close kinetic chain exercises — CKC include mini squats, leg press, step-up and step-down, wall slides etc along with their respective modality as quadriceps drill and static cycle ergometer respectively on grade-3 knee OA patients
  Arms: Group A: close kinetic chain exercises
Other: open kinetic chain exercises — The distal segment of the body components can move freely during OKC exercise.OKC exercises include quadriceps setting, knee extension in sitting and straight leg raise in lying position; it also includes quadriceps drills as part of OKC exercises
  Arms: Group B: open kinetic chain exercises

SUMMARY:
A randomized clinical trial will be conducted in Gujranwala and 24 patients with grade 3 knee OA will be recruited. After consent, patients will be randomly allocated into 2 groups by lottery method. Group A will do close kinetic chain exercises, including static cycling, lifestyle modification, and patient education. Group B will do open kinetic chain exercises including quadriceps drills with lifestyle modification and patient education. A total duration of 12 weeks with 3 sessions per week will be given. Outcome measures Assessment will be done at 0 weeks, 4 weeks, 8 weeks, and 12 weeks.

DETAILED DESCRIPTION:
Osteoarthritis is a clinical syndrome characterized by joint pain, varying degrees of functional impairment, and a poor quality of life and in 21st century It is predicted that the number of persons over 65 would double placing a heavy burden on healthcare systems and caregivers' resources. For individuals with knee OA, open kinetic chain (OKC) and closed kinetic chain (CKC) exercises have been recommended thus far. The distal segment of the body components can move freely during OKC exercise since it is not bound, but remain static on the ground during CKC exercise.

A single-blinded randomized clinical trial will be conducted at Al-Raee Trust Hospital Gujranwala and 24 patients of both genders and age of 50-70 years with grade 3 knee OA (according to Kellgren and Lawrence classification system based on plain x-rays) will be recruited. After taking written consent, patients will be randomly allocated into 2 groups by lottery method. Group A will be treated with close kinetic chain exercises including static cycling with lifestyle modification and patient's education and group B will be treated with open kinetic chain exercises including quadriceps drill with lifestyle modification and patient's education about 30 minutes per session including 10 min of walking as a warm up for total duration of 12 weeks with 3 sessions per week. Outcome measures such as pain, disability and health status will be assessed by NPRS, WOMAC and OAKHQOL respectively. Assessment will be done by therapist at 0 week, 4 weeks, 8 weeks and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* • Both genders

  * With Grade 3 of Knee Osteoarthritis (Kellgren-Lawrence scoring)
  * Mild-to-moderate pain on NPRS
  * Age 50-70 years old
  * Available three times a week for over 3 months

Exclusion Criteria:

* • Having Knee surgery in the past 6 months

  * Having Acute symptomatic KOA
  * Having Any muscular, joint or neurological conditions that affect lower limb function
  * Conducting another structured exercise programme specifically for KOA during this study period
  * Having Motor neuron disorders such as Alzheimer's and Parkinson's diseases.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale: | up to 12 weeks
  Pain intensity will be assessed by NPRS. The 11-point NPRS (intervals from 0-10) is used to quantify pain intensity; 0 represents no pain, and 10 represent the worst possible agony. The NPRS is an valid and reliable instrument for older persons. Participants will be asked to select the number that most accurately describes their level of pain. At the baseline assessment, following each exercise session during the 12-week intervention, and finally at the end of the intervention programme, the NPRS scores will be recorded
Western Ontario and McMaster Universities Arthritis Index | up to 12 weeks
  This questionnaire is designed to evaluate an osteoarthritis patient's level of disability. It consists of 24 items that assess the patient's health and function in a variety of ways, including: clinical symptoms (5 questions), the severity of joint stiffness (2 questions), and daily living activities (17 questions). There are five subscales for each question, with the best situation scoring as never or none and the worst situation scoring as extreme or always. Higher ratings in this case indicate a better position and less suffering. Scores will be recorded after each session of intervention at 0 week, 4 weeks, 8 weeks and 12 weeks
Osteoarthritis Knee and Hip Quality of Life Score | up to 12 weeks
  The Osteoarthritis Knee and Hip Quality of Life (OAKHQOL) was created to assess patients with hip and knee OA's quality of life particularly. The OAKHQOL is a reliable and valid tool for measuring the health-related quality of life of people with knee OA. Physical activities (16 items), mental health (13 items), pain (4 items), social support (4 items), social functioning (3 items), and 3 independent items are among the 43 items that make up the OAKHQOL questionnaire, which describes quality of life in five domains. Each item is graded from 0 to 10 on a scale. The mean of all the components constitutes the final score. The sum of all the mean scores will result in a scale from 0 (the highest achievable QOL) to 100 (worst possible QOL)

CONTACTS AND LOCATIONS:
Overall Officials: Rida Shakeel, MS*, Principal Investigator — Riphah International University
Locations (1):
- Al-Raee Trust Hospital, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Raposo F, Ramos M, Lucia Cruz A. Effects of exercise on knee osteoarthritis: A systematic review. Musculoskeletal Care. 2021 Dec;19(4):399-435. doi: 10.1002/msc.1538. Epub 2021 Mar 5. PMID 33666347
- [Background] Primorac D, Molnar V, Rod E, Jelec Z, Cukelj F, Matisic V, Vrdoljak T, Hudetz D, Hajsok H, Boric I. Knee Osteoarthritis: A Review of Pathogenesis and State-Of-The-Art Non-Operative Therapeutic Considerations. Genes (Basel). 2020 Jul 26;11(8):854. doi: 10.3390/genes11080854. PMID 32722615
- [Background] Olagbegi OM, Adegoke BO, Odole AC. Effectiveness of three modes of kinetic-chain exercises on quadriceps muscle strength and thigh girth among individuals with knee osteoarthritis. Arch Physiother. 2017 Jul 19;7:9. doi: 10.1186/s40945-017-0036-6. eCollection 2017. PMID 29340203
- [Background] Luan L, Bousie J, Pranata A, Adams R, Han J. Stationary cycling exercise for knee osteoarthritis: A systematic review and meta-analysis. Clin Rehabil. 2021 Apr;35(4):522-533. doi: 10.1177/0269215520971795. Epub 2020 Nov 10. PMID 33167714
- [Background] Sanchez Romero EA, Fernandez Carnero J, Villafane JH, Calvo-Lobo C, Ochoa Saez V, Burgos Caballero V, Laguarta Val S, Pedersini P, Pecos Martin D. Prevalence of Myofascial Trigger Points in Patients with Mild to Moderate Painful Knee Osteoarthritis: A Secondary Analysis. J Clin Med. 2020 Aug 7;9(8):2561. doi: 10.3390/jcm9082561. PMID 32784592
- [Background] Ng WH, Jamaludin NI, Sahabuddin FNA, Ab Rahman S, Ahmed Shokri A, Shaharudin S. Comparison of the open kinetic chain and closed kinetic chain strengthening exercises on pain perception and lower limb biomechanics of patients with mild knee osteoarthritis: a randomized controlled trial protocol. Trials. 2022 Apr 15;23(1):315. doi: 10.1186/s13063-022-06153-8. PMID 35428274
- [Background] Goetz C, Ecosse E, Rat AC, Pouchot J, Coste J, Guillemin F. Measurement properties of the osteoarthritis of knee and hip quality of life OAKHQOL questionnaire: an item response theory analysis. Rheumatology (Oxford). 2011 Mar;50(3):500-5. doi: 10.1093/rheumatology/keq357. Epub 2010 Nov 11. PMID 21071480